CLINICAL TRIAL: NCT04602546
Title: Evaluation of BIS™ and Levels of Sedation With Common Inhalational Anesthetics in Healthy Volunteers (OLIVER)
Brief Title: Evaluation of Bispectral Index (BIS™) and Levels of Sedation With Common Inhalational Anesthetics in Healthy Volunteers (OLIVER)
Acronym: OLIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MDT19053OLIVER
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized study to collect data to evaluate the relationship between BIS and inhaled anesthetics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Sevoflurane alone (Active Comparator): Sevoflurane will be administered in steps to achieve a loss of consciousness via a tight-face mask by increasing the end-tidal concentration of Sevoflurane (ETSEVO). Targeted concentration for ETSEVO are 0.25, 0.5, 0.75, 1, 3, 4, 5% or higher until MOAA/S scales at values less than 2 is reached.
  The equilibration time for each targeted concentration will be approximately 12 minutes to maintain a constant ETSEVO. The BIS™ value, MOAA/S score and picture recall test will be assessed when the patient is awake and at the different ETSEVO concentrations.
  ETSEVO is decreased by the same steps until consciousness is regained.
  Interventions: Device: BIS Complete Monitoring System
- Sevoflurane with Remifentanil Group (Active Comparator): Two (2) minutes before starting sevoflurane, to attain an effect-site targeted concentration of remifentanil of 4 ng/ml, an initial IV bolus of remifentanil will be given followed by the start of an infusion. Approximately within 7 minutes, the infusion rate of remifentanil may be adjusted to maintain the effect-site concentration of remifentanil of 4 ng/ml.
  Sevoflurane will be administered via a tight-face mask in steps to achieve a loss of consciousness by increasing the end-tidal concentration of Sevoflurane (ETSEVO). Targeted concentration for ETSEVO are 0.25, 0.5, 0.75, 1, 3, 4, 5% or higher until an MOAA/S score of less than 2 is reached.
  ETSEVO is decreased by the same steps until consciousness is regained.
  Interventions: Device: BIS Complete Monitoring System
- Sevoflurane with Fentanyl Group (Active Comparator): Two (2) minutes before starting sevoflurane, to attain an effect-site targeted concentration of fentanyl of 2 ng/mL, an initial IV bolus of fentanyl will be given followed by the start of an infusion. Approximately within 10 minutes, the infusion rate of fentanyl may be adjusted to maintain the effect-site concentration of fentanyl of 2 ng/ml.
  Sevoflurane will be administered via a tight-face mask in steps to achieve a loss of consciousness by increasing the end-tidal concentration of Sevoflurane (ETSEVO). Targeted concentration for ETSEVO are 0.25, 0.5, 0.75, 1, 3, 4, 5% or higher until an MOAA/S score of equal to or less than 2 is reached.
  ETSEVO is decreased by the same steps until consciousness is regained.
  Interventions: Device: BIS Complete Monitoring System
- Desflurane Group (Active Comparator): Due to desflurane being a volatile agent and not well tolerated as an induction agent, an initial IV bolus of 1% propofol provided at 2mg/kg, with supplemental boluses given at the investigators discretion in order to achieve laryngeal mask (LMA) insertion, will be administered 15-20 minutes prior to desflurane. Once correct LMA placement has been confirmed, there will be an equilibrium time of approximately 15-20 minutes to allow the effect site concentration of propofol to reach a level consistent with a pharmacodynamic effect of consciousness as measured by a MOAA/S score of 2 or 3. Desflurane will then be administered via a tight-face mask at the targeted end-tidal concentration (ETDES) of 2, 5, 7, 8, 9, 10 %, or higher until an MOAA/S score of less than 2 is reached.
  The BIS™ value will be correlated with desflurane ETDES concentration. ETDES is decreased by the same steps until consciousness is regained.
  Interventions: Device: BIS Complete Monitoring System
- Isoflurane Group (Active Comparator): Due to isoflurane being a volatile agent and not well tolerated as an induction agent, an initial IV bolus of 1% propofol provided at 2mg/kg, with supplemental boluses given at the investigators discretion in order to achieve LMA insertion, will be administered 15-20 minutes prior to isoflurane.Isoflurane will be administered via a tight-face mask in steps to achieve a loss of consciousness (MOAA/S of 0,1) by increasing the end-tidal concentration of Isoflurane (ETISO). Targeted concentration for ETISO are 0.25, 0.5, 0.75, 1, 1.5% or higher until MOAA/S scales at values less than 2 is reached.
  The BIS™ value will be correlated with desflurane ETISO concentration. ETISO is decreased by the same steps until consciousness is regained.
  Interventions: Device: BIS Complete Monitoring System

INTERVENTIONS:
Device: BIS Complete Monitoring System — The BIS™ EEG complete monitoring system is intended for use under the direct supervision of a licensed healthcare practitioner or by personnel trained in its proper use. The system and its associated parameters are intended for use on adult patients within a hospital or medical facility, providing patient care to monitor the state of the brain by data acquisition of EEG signals.

SUMMARY:
To investigate the relationship between BIS™ and inhaled anesthetics across a wide range of anesthetic concentration and hypnotic states, and to provide evidence to support BIS™ performance in use with Isoflurane, Sevoflurane and Desflurane in combination with opioids.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (ASA physical status 1), male or female subjects between the ages of 18 to 60 years;
2. Completion of a health screening for a medical history by a licensed physician, nurse practitioner or physician assistant;
3. Vital signs must be within the following ranges to be included: Vital signs measured sitting after 3 minutes rest; heart rate: 45-90 bpm; systolic blood pressure: 110-140; diastolic blood pressure: 50-90. Out-of-range vital signs may be repeated once. [Pre-dose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified sub-investigator) before study drug administration. The Principal Investigator or designee will verify the eligibility of each subject with out-of-range vital signs and document approval before dosing].

Exclusion Criteria:

1. Has severe contact allergies that may cause a reaction to standard adhesive materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes, or other medical sensors [self-reported];
2. Known neurological disorder (e.g., epilepsy, the presence of a brain tumor, a history of brain surgery, hydrocephalic disorders, depression needing treatment with anti-depressive drugs, a history of brain trauma) [self-reported and assessment by PI or delegate];
3. Known cardiovascular disease (e.g., hypertension, coronary artery disease, prior acute myocardial infarction, any valvular and/or myocardial disease involving a decrease in ejection fraction, arrhythmias, which are either symptomatic or require continuous medication/ pacemaker/ automatic internal cardioverter defibrillator), current implanted pacemaker or automatic internal cardioverter defibrillator [self-reported and assessment by PI or delegate];
4. Has a clinically significant abnormal finding on medical history, physical examination, clinical laboratory tests, or ECG at the screening [self-reported and assessment by PI or delegate];
5. Use of psychoactive medication within the past 60 days (e.g., benzodiazepines, antiepileptic drugs, Parkinson's medication, anti-depressant drugs, opioids) [self-reported and assessment by PI or delegate];
6. Subjects with known gastric diseases [self-reported and assessment by PI or delegate];
7. Has a positive urine cotinine test or urine drug screen or oral ethanol test [Point of Care (POC) testing];
8. Known history of allergic or adverse response to drugs to be administered [self-reported];
9. Known history of complications relating to previous general anesthesia or conscious sedation [self-reported and assessment by PI or delegate];
10. Known history of malignant hyperthermia [self-reported and assessment by PI or delegate];
11. Has a room air saturation less than 95% by pulse oximetry [measurement by PI or delegate];
12. Has a clinically significant abnormal pulmonary function test via spirometry [assessment by PI or delegate];
13. Pregnant or lactating women [assessed by urine test and self-reported];
14. Subjects with tattooed skin specific to the sensor placement areas (forehead, fingers, chest) [self-reported and assessment by PI or delegate];
15. The subject must not take any prescription medication, except female hormonal contraceptives or hormone replacement therapy, from 14 days before the dosing until the end-of-study visit without evaluation and approval by the Investigator. Subjects who participated in a previous clinical trial who received a required FDA approved concomitant medication, for example, naltrexone, but were not randomized may be considered for participation in this study if they meet the washout requirement [assessment by PI or delegate].

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David MacLeod, MBBS, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - University of California at San Francisco, San Francisco, California
  - Duke University Medical Center, Durham, North Carolina
  - University of Utah Health Science Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects without a procedure (n=49) include screen failure (n=14), withdrawal by subject (n=11), informed consent passed 60 day limit (n=18), physician decision (n=1), sponsor request (n=2), and other (n=3)
Groups:
- Sevoflurane Alone: Sevoflurane will be administered in steps to achieve a loss of consciousness via a tight-face mask by increasing the end-tidal concentration of Sevoflurane (ETSEVO). Targeted concentration for ETSEVO are 0.25, 0.5, 0.75, 1, 3, 4, 5% or higher until MOAA/S scales at values less than 2 is reached.
  The equilibration time for each targeted concentration will be approximately 12 minutes to maintain a constant ETSEVO. The BIS™ value, MOAA/S score and picture recall test will be assessed when the patient is awake and at the different ETSEVO concentrations.
  ETSEVO is decreased by the same steps until consciousness is regained.
  BIS Complete Monitoring System: The BIS™ EEG complete monitoring system is intended for use under the direct supervision of a licensed healthcare practitioner or by personnel trained in its proper use. The system and its associated parameters are intended for use on adult patients within a hospital or medical facility, providing patient care to monitor the state of the brain by data acquisition of EEG signals.
- Sevoflurane With Remifentanil Group: Two (2) minutes before starting sevoflurane, to attain an effect-site targeted concentration of remifentanil of 4 ng/ml, an initial IV bolus of remifentanil will be given followed by the start of an infusion. Approximately within 7 minutes, the infusion rate of remifentanil may be adjusted to maintain the effect-site concentration of remifentanil of 4 ng/ml.
  Sevoflurane will be administered via a tight-face mask in steps to achieve a loss of consciousness by increasing the end-tidal concentration of Sevoflurane (ETSEVO). Targeted concentration for ETSEVO are 0.25, 0.5, 0.75, 1, 3, 4, 5% or higher until an MOAA/S score of less than 2 is reached.
  ETSEVO is decreased by the same steps until consciousness is regained.
  BIS Complete Monitoring System: The BIS™ EEG complete monitoring system is intended for use under the direct supervision of a licensed healthcare practitioner or by personnel trained in its proper use. The system and its associated parameters are intended for use on adult patients within a hospital or medical facility, providing patient care to monitor the state of the brain by data acquisition of EEG signals.
- Sevoflurane With Fentanyl Group: Two (2) minutes before starting sevoflurane, to attain an effect-site targeted concentration of fentanyl of 2 ng/mL, an initial IV bolus of fentanyl will be given followed by the start of an infusion. Approximately within 10 minutes, the infusion rate of fentanyl may be adjusted to maintain the effect-site concentration of fentanyl of 2 ng/ml.
  Sevoflurane will be administered via a tight-face mask in steps to achieve a loss of consciousness by increasing the end-tidal concentration of Sevoflurane (ETSEVO). Targeted concentration for ETSEVO are 0.25, 0.5, 0.75, 1, 3, 4, 5% or higher until an MOAA/S score of equal to or less than 2 is reached.
  ETSEVO is decreased by the same steps until consciousness is regained.
  BIS Complete Monitoring System: The BIS™ EEG complete monitoring system is intended for use under the direct supervision of a licensed healthcare practitioner or by personnel trained in its proper use. The system and its associated parameters are intended for use on adult patients within a hospital or medical facility, providing patient care to monitor the state of the brain by data acquisition of EEG signals.
- Desflurane Group: Due to desflurane being a volatile agent and not well tolerated as an induction agent, an initial IV bolus of 1% propofol provided at 2mg/kg, with supplemental boluses given at the investigators discretion in order to achieve LMA insertion, will be administered 15-20 minutes prior to desflurane. Once correct LMA placement has been confirmed, there will be an equilibrium time of approximately 15-20 minutes to allow the effect site concentration of propofol to reach a level consistent with a pharmacodynamic effect of consciousness as measured by a MOAA/S score of 2 or 3. Desflurane will then be administered via a tight-face mask at the targeted end-tidal concentration (ETDES) of 2, 5, 7, 8, 9, 10 %, or higher until an MOAA/S score of less than 2 is reached.
  The BIS™ value will be correlated with desflurane ETDES concentration. ETDES is decreased by the same steps until consciousness is regained.
  BIS Complete Monitoring System: The BIS™ EEG complete monitoring system is intended for use under the direct supervision of a licensed healthcare practitioner or by personnel trained in its proper use. The system and its associated parameters are intended for use on adult patients within a hospital or medical facility, providing patient care to monitor the state of the brain by data acquisition of EEG signals.
- Isoflurane Group: Due to isoflurane being a volatile agent and not well tolerated as an induction agent, an initial IV bolus of 1% propofol provided at 2mg/kg, with supplemental boluses given at the investigators discretion in order to achieve LMA insertion, will be administered 15-20 minutes prior to isoflurane.Isoflurane will be administered via a tight-face mask in steps to achieve a loss of consciousness (MOAA/S of 0,1) by increasing the end-tidal concentration of Isoflurane (ETISO). Targeted concentration for ETISO are 0.25, 0.5, 0.75, 1, 1.5% or higher until MOAA/S scales at values less than 2 is reached.
  The BIS™ value will be correlated with desflurane ETISO concentration. ETISO is decreased by the same steps until consciousness is regained.
  BIS Complete Monitoring System: The BIS™ EEG complete monitoring system is intended for use under the direct supervision of a licensed healthcare practitioner or by personnel trained in its proper use. The system and its associated parameters are intended for use on adult patients within a hospital or medical facility, providing patient care to monitor the state of the brain by data acquisition of EEG signals.
Period: Overall Study
Arm/Group | Sevoflurane Alone | Sevoflurane With Remifentanil Group | Sevoflurane With Fentanyl Group | Desflurane Group | Isoflurane Group
Started | 33 | 29 | 32 | 35 | 33
Completed | 29 | 27 | 29 | 28 | 30
Not Completed | 4 | 2 | 3 | 7 | 3
Not completed — Training | 2 | 2 | 1 | 2 | 0
Not completed — Randomized with disqualified data | 2 | 0 | 2 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sevoflurane Alone | Sevoflurane With Remifentanil Group | Sevoflurane With Fentanyl Group | Desflurane Group | Isoflurane Group | Total
Number analyzed (Participants) | 29 | 27 | 29 | 28 | 30 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (8.4) | 25.7 (4.6) | 24.1 (4.5) | 28.6 (7.9) | 25.4 (6.1) | 26.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 13 | 16 | 14 | 69
  Male | 18 | 12 | 16 | 12 | 16 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 5 | 8 | 3 | 27
  Not Hispanic or Latino | 24 | 21 | 22 | 20 | 27 | 114
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 0 | 0 | 3
  Asian | 5 | 9 | 9 | 2 | 6 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 2 | 2 | 2 | 6 | 19
  White | 14 | 14 | 16 | 20 | 16 | 80
  More than one race | 1 | 1 | 0 | 3 | 0 | 5
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 29 | 27 | 29 | 28 | 30 | 143

OUTCOME MEASURES:

1. Primary Outcome: BIS 50
Description: To determine BIS50, the BIS™ value (index score on a scale of 0-100 (0 being dead and 100 being fully awake/responsive) on the BIS™ monitor) at which 50% of patients will be unresponsive at a given drug concentration. Responsiveness is measured using the Modified Observer's Assessment of Alertness and Sedation (MOAAS) a 0-5 scale where 0 represents no response to deep stimulus and 5 represents fully awake).
Time Frame: duration of anesthesia administration, up to 2 hours
Measure: Mean (95% Confidence Interval); unit: units on a scale 0-100
Arm/Group | Sevoflurane Alone | Sevoflurane With Remifentanil Group | Sevoflurane With Fentanyl Group | Desflurane Group | Isoflurane Group
Number analyzed (Participants) | 29 | 27 | 29 | 28 | 30
units on a scale 0-100 | 72.3 [70.1 to 74.3] | 74.2 [72.6 to 75.7] | 76.2 [74.3 to 78.0] | 67.5 [63.5 to 71.7] | 72.2 [69.5 to 74.8]

2. Secondary Outcome: BIS 95
Description: To determine BIS95, the BIS™ value (index score on a scale of 0-100 (0 being dead and 100 being fully awake/responsive) on the BIS™ monitor) at which 95% of patients will be unresponsive at a given drug concentration. Responsiveness is measured using the Modified Observer's Assessment of Alertness and Sedation (MOAAS) a 0-5 scale where 0 represents no response to deep stimulus and 5 represents fully awake).
Time Frame: duration of anesthesia administration
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Sevoflurane Alone | Sevoflurane With Remifentanil Group | Sevoflurane With Fentanyl Group | Desflurane Group | Isoflurane Group
Number analyzed (Participants) | 29 | 27 | 29 | 28 | 30
units on a scale | 58.4 [52.9 to 61.9] | 62.3 [58.5 to 64.9] | 60.6 [55.8 to 63.9] | 49.1 [41.0 to 54.3] | 54.8 [48.2 to 59.2]

3. Secondary Outcome: Prediction Probability (PK)
Description: To determine if the value on the BIS™ monitor (index score on a scale of 0-100 (0 being dead and 100 being fully awake/responsive) on the BIS™ monitor) can predict the subject's responsiveness at a given drug concentration. Responsiveness is measured using the Modified Observer's Assessment of Alertness and Sedation (MOAAS) a 0-5 scale where 0 represents no response to deep stimulus and 5 represents fully awake).
Time Frame: duration of anesthesia administration, up to 2 hours
Measure: Mean (95% Confidence Interval); unit: Prediction Probability
Arm/Group | Sevoflurane Alone | Sevoflurane With Remifentanil Group | Sevoflurane With Fentanyl Group | Desflurane Group | Isoflurane Group
Number analyzed (Participants) | 29 | 27 | 29 | 28 | 30
Prediction Probability | 0.967 [0.951 to 0.983] | 0.960 [0.942 to 0.979] | 0.945 [0.924 to 0.967] | 0.977 [0.960 to 0.995] | 0.957 [0.934 to 0.980]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from enrollment through study exit, up to 48 hours
Arm/Group | Sevoflurane Alone | Sevoflurane With Remifentanil Group | Sevoflurane With Fentanyl Group | Desflurane Group | Isoflurane Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29 | 0/32 | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/29 | 0/32 | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 13/33 | 24/29 | 29/32 | 14/35 | 18/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sevoflurane Alone (N=33) | Sevoflurane With Remifentanil Group (N=29) | Sevoflurane With Fentanyl Group (N=32) | Desflurane Group (N=35) | Isoflurane Group (N=33)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 15 (15) | 2 (2) | 7 (7) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 12 (12) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 5 (5) | 8 (8) | 8 (8) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5) | 13 (13) | 21 (21) | 3 (3) | 9 (9)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT04602546/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT04602546/SAP_001.pdf